CLINICAL TRIAL: NCT04040504
Title: Clinical Efficacy and Infection Risk of ERCP Using a Novel Duodenoscope With a Disposable Cap: a Randomized Controlled Trial
Brief Title: Infection Control in ERCP Using a Duodenoscope With a Disposable Cap
Acronym: ICECAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Nauzer Forbes, Clinical Assistant Professor of Medicine, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB19-0983
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Bile Duct Diseases
MeSH Terms: conditions — Bile Duct Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient, investigator and outcomes assessors will be blinded to the intervention. The endoscopist will not be blinded, since the type of scope and cap being used can be detected during the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentax ED-34i10T2 Duodenoscope with Disposable Cap (DEC) (Experimental): Pentax ED-34i10T2 Duodenoscope with Disposable Cap (DEC)
  Interventions: Device: ERCP procedure with Pentax ED-34i10T2 Duodenoscope with Disposable Cap (DEC)
- Pentax ED-34i10T Duodenoscope (Active Comparator): Pentax ED-34i10T Duodenoscope
  Interventions: Device: ERCP procedure with Pentax ED-34i10T Duodenoscope

INTERVENTIONS:
Device: ERCP procedure with Pentax ED-34i10T2 Duodenoscope with Disposable Cap (DEC) — ERCP procedure using Pentax ED-34i10T2 Duodenoscope with Disposable Cap (DEC) and any necessary accessories.
  Arms: Pentax ED-34i10T2 Duodenoscope with Disposable Cap (DEC)
Device: ERCP procedure with Pentax ED-34i10T Duodenoscope — ERCP procedure using Pentax ED-34i10T Duodenoscope with any necessary accessories.
  Arms: Pentax ED-34i10T Duodenoscope

SUMMARY:
1. Background & Rationale

   Over 650,000 endoscopic retrograde cholangio-pancreatography (ERCP) procedures are performed annually in the United States alone. ERCP is universally performed using a highly specialized type of flexible endoscope called a duodenoscope. Though critical for the successful completion of ERCP, the design of duodenoscopes makes them among the most complicated medical devices that require routine disinfection and reprocessing. In recent years, several ERCP-related infectious outbreaks have occurred.

   Thus, it is clear that novel strategies need to be developed in order to prevent future ERCP-related outbreaks. Specialized duodenoscopes with disposable caps have been developed, and these represent a promising new modality with the potential to drastically reduce the rates of duodenoscope-related infection.
2. Research Questions & Objectives

   There are two co-primary outcomes in this study; the first is to determine the clinical efficacy of a novel duodenoscope with a disposable elevator cap (DEC) system compared with a duodenoscope with a traditional design. The second co-primary objective is to determine the rate of persistent pathogenic contamination of the novel duodenoscope following standardized disinfection and reprocessing protocols compared with a traditional duodenoscope.
3. Methods

This is a prospective, consecutive, randomized controlled study. The intervention arm will comprise use of the ED34-i10T2 duodenoscope with DEC, along with any required standard ERCP accessories, whereas the control arm will comprise use of the ED34-i10T duodenoscope with any required ERCP accessories. All procedures will be performed by expert endoscopists with adequate training, or by advanced endoscopy trainees under direct supervision.

Collected data will include primary endpoints listed above, in addition to patient demographics, endoscopist and trainee data, sedation used, procedural details, and peri-procedural data. Data will be collected at index procedure and at 30-day follow-up. All data will be recorded on REDCap.

DETAILED DESCRIPTION:
There are two co-primary objectives of this study; the first is to determine the clinical efficacy of a novel duodenoscope with a disposable elevator cap (DECTM) system compared with a duodenoscope with a traditional design. The second is to determine the rate of persistent pathogenic contamination of the novel duodenoscope following standardized disinfection and reprocessing protocols, compared with a traditional duodenoscope.

This is a prospective, consecutive, randomized controlled study which will assess 1) the clinical efficacy of DEC versus standard duodenoscopes and 2) the persistent bacterial contamination rate of DEC versus standard duodenoscopes. The intervention arm will comprise use of the ED34-i10T2 duodenoscope with DEC, along with any required standard ERCP accessories, whereas the control arm will comprise use of the ED34-i10T duodenoscope with any required ERCP accessories. The study will take place at a single high-volume tertiary ERCP referral center in Calgary, Alberta, Canada, where over 1,500 ERCPs are performed annually. All procedures will be performed by trained endoscopists having each performed over 1,000 ERCPs or by advanced therapeutic endoscopy trainees under direct supervision of the expert endoscopists.

All consecutive patients at the study center who meet the eligibility criteria below will be invited for participation in the study. Patients who sign the informed consent form will be considered enrolled. In cases where it is determined that the patient failed to meet the eligibility criteria after the patient has agreed to participate in the study and/or has signed the informed consent, the study personnel will complete screening forms as well as indicate the specific inclusion/exclusion criterion that was not met. Such a patient will be considered a screen failure and will not count towards the final analyses.

Patients fulfilling the inclusion/exclusion criteria above will be randomized following consent in a 1:1 ratio. Permuted block randomization will be utilized in blocks of 8 patients. Allocation will be to one of two groups: 1) ERCP using ED34-i10T2 duodenoscope with DEC or 2) ERCP using a conventional duodenoscope (ED34-i10T). Confidential random number allocation will be accessed via a secure internet software. The study investigators, outcome adjudicators and patients will be blinded to allocation. The endoscopist will not be blinded. In cases where additional or alternate duodenoscope(s) is/are required to achieve the desired goal of the ERCP procedure, the choice(s) of device(s) will be left to the discretion of the endoscopist, regardless of the study arm to which the patient has been allocated.

The investigators have previously designed and implemented the Calgary Registry for Advanced and Therapeutic Endoscopy (CReATE, University of Calgary Conjoint Health Research Ethics Board 18-0410). CReATE is a high-fidelity prospective database that seeks to answer questions in ERCP outcomes research. As such, over 400 data fields are collected in real-time for each ERCP procedure, including detailed patient-, endoscopist- and procedure-based variables. Therefore, CReATE serves as the ideal data collection platform for this prospective randomized trial.

Data are inputted by a full-time research assistant, and stored and managed on a secure web application specializing in healthcare database implementation and maintenance, REDCap.19 This web portal allows for facile access to secure data. The web portal is secured by the latest security technology. Study participants will be identifiable on the secure platform for purposes of patient contact, follow-up and potential withdrawal. For the purposes of this randomized study, an additional tab will be created in the electronic interface that will allow for entry of the arm to which the patient has been randomized. Whenever data are exported for analysis, they will be de-identified and assigned unique study codes only. The primary investigator will be the custodian of the identifiable electronic data, which will be stored only on a secure server accessible only via combination of password protection and temporary electronic fob.

Consecutive patients undergoing ERCP will be flagged as potentially eligible for study participation. On the day of the procedure, the patient will be approached by a research assistant (RA), who will explain the study, confirm eligibility, and answer any potential questions. If the patient agrees to participate, the relevant informed consent form is signed and witnessed. If the patient decides not to participate, the ERCP proceeds as per the usual standard of care, with or without the use of DEC as per the endoscopist's discretion (and the sequence that follows does not apply).

1. The RA collects any relevant patient-related and pre-procedural data through combination of direct patient interview and review of the medical records.
2. The patient is randomized to one of the two study arms.
3. The patient enters the endoscopy/fluoroscopy room and the procedure commences.
4. During the ERCP procedure, relevant peri-procedural data are recorded by the RA by direct observation, and/or, if necessary, in consultation with the procedural physician(s) and/or nurse(s).
5. After the procedure is complete, the patient is moved to the recovery room for observation. Depending on their disposition and the course of the procedure, observation times and protocols differ. During this stage, the RA collects any relevant post-procedural data, and any missing pre- or peri-procedural data.
6. Any peri- or immediate post-procedural adverse event(s) is/are recorded.
7. The patient is examined by the endoscopist prior to discharge and provided with written post-procedure information, including a phone number to call in the event of any issues.
8. The RA meets with the patient prior to their discharge from the unit to answer any final potential questions.

After the ERCP is complete, the in-room nursing team will carry out standardized post-endoscopy manual cleaning and disinfection of the DEC or traditional duodenoscope. In cases where the DEC was used, the cap will be disposed of. These processes will be timed by the research assistant. Following this, the scope will be portered to the automated reprocessing room for disinfection and reprocessing, which will also be timed.

After reprocessing, staff will then observe the following sequence to determine whether there is any persistent bacterial contamination despite standardized disinfection and reprocessing. These samples will then be shipped for microbiologic analysis. The protocol for duodenoscope sampling that will be utilized for this study is adapted from the Duodenoscope Surveillance Sampling and Culturing Protocols, which were developed jointly by the Department of Health and Human Services, Food and Drug Administration (FDA), Centers for Disease Control and Prevention (CDC), and American Society for Microbiology (ASM).24 The procedure is summarized here.

1. Two staff are needed to conduct sampling from duodenoscope channels; one person (the sampler) will maintain aseptic handling and conduct brushing steps, while the second person (the facilitator) will open packages and handle the unsampled portions of the duodenoscope.
2. The staff will label the sterile sample containers with relevant information.
3. The staff will don their personal protective equipment (PPE).
4. The staff will set the duodenoscope on a sterile drape.
5. Two samples will be collected and combined. First, an instrument channel sample (from the biopsy port to the distal scope end) will be taken.
6. Second, an elevator recess sample will be taken by flushing and brushing of the elevator recess (in the case of the disposable cap, the distal scope tip to which the disposable cap attaches will be sampled instead, ensuring sampling of the joint line between cap and scope).
7. The duodenoscope will then be handled and transported back to the endoscopy unit according to our local institutional policies.
8. Samples will be packed in appropriate biohazard containers, packaged, and transported for microbiologic analysis. The samples will be assigned a unique study number so that the microbiologic analysts will be blinded to the type of duodenoscope that was used for the index procedure.

The presence of any post-reprocessing bacterial population(s) will be assessed using plating for growth aerobic and anaerobic conditions. If after 72 hours there is no growth, the sample will be deemed negative, and will be discarded. Positive samples will further be characterized using serial dilutions to establish colony-forming unit (CFU) counts and sequenced for characterization of bacterial communities using a 16S rRNA amplicon Next-generation sequencing (NGS).

Patients will be contacted by the RA by telephone 30 days following their ERCP to assess for any ongoing symptoms and advise of any adverse events, including unplanned emergency department visits or inpatient admissions. The patient's medical record is also reviewed at 30 days for complete details of any unplanned emergency department visits, inpatient admissions or prolonged admissions.

In accordance with the Declaration of Helsinki and the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use Good Practice Guidelines, a participant is free to withdraw from participation in the study at any time, for any reason without prejudice to their future medical care by the physician or the institution. The investigator(s) may also withdraw the participant at any time in the interests of patient safety. Participants may be removed from the study if one or more of the following events occur:

* withdrawal of consent;
* decision is made by the investigator(s) that removal from the study is in the patient's best medical interest;
* study is stopped by ethics/regulatory authorities.

If a subject withdraws from the clinical investigation, the primary or any additional reason(s) shall be reported. All applicable case report forms up to the point of subject withdrawal, including an End of Study form, should be completed.

Subjects who are "lost-to-follow-up" will have three documented attempts to contact them prior to completion of the End of Study form. If withdrawal is due to investigator's discretion, the investigator should describe what follow-up activities the investigator shall perform. Unless the withdrawal is due to a Serious Adverse Event (SAE), additional subject data will not be collected after the point at which the subject has been withdrawn or withdraws consent from the study. Data collected up to the point of withdrawal may be used by the investigators as permitted in the Informed Consent Form (ICF).

This clinical trial will be considered complete when participants are no longer being examined or the last participant's final 30-day follow-up check has occurred. A participant will be considered to have completed the study if he or she has completed the index procedure in addition to the follow-up phone assessment at the 30-day timepoint.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or over;
* ability to give informed consent to involvement;
* requirement for ERCP to be performed for any indication.

Exclusion Criteria:

* age < 18 years;
* inability or unwillingness to provide informed consent;
* standard contraindications to ERCP;
* pregnant status or breastfeeding mother;
* inability to successfully complete procedure under conscious sedation;
* out-of-province status;
* incarceration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
ERCP technical success rate | Immediate
  Technical success will be determined in duplicate by two blinded outcome adjudicators with no knowledge of the patient's allocation in the study. The adjudicators will review redacted and de-identified procedure reports for each study patient, and determine the presence or absence of technical success of the overall procedure based on a set of a priori definitions.
Persistent bacterial contamination rate | Immediate
  Persistent bacterial contamination will be assessed following standardized disinfection and reprocessing using microbiologic swabs and culturing.

CONTACTS AND LOCATIONS:
Overall Officials: Nauzer Forbes, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- Peter Lougheed Centre, Calgary, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Forbes N, Elmunzer BJ, Allain T, Parkins MD, Sheth PM, Waddell BJ, Du K, Douchant K, Oladipo O, Saleem A, Cartwright S, Chau M, Howarth M, McKay J, Nashad T, Ruan Y, Bishay K, Gonzalez-Moreno E, Meng ZW, Bass S, Bechara R, Cole MJ, Jalink DW, Mohamed R, Turbide C, Belletrutti PJ, Kayal A, Kumar PR, Hilsden RJ, Buret AG, Hookey L, Heitman SJ. Effect of Disposable Elevator Cap Duodenoscopes on Persistent Microbial Contamination and Technical Performance of Endoscopic Retrograde Cholangiopancreatography: The ICECAP Randomized Clinical Trial. JAMA Intern Med. 2023 Mar 1;183(3):191-200. doi: 10.1001/jamainternmed.2022.6394. PMID 36689215
- [Derived] Forbes N, Elmunzer BJ, Allain T, Chau M, Koury HF, Bass S, Belletrutti PJ, Cole MJ, Gonzalez-Moreno E, Kayal A, Kumar P, Mohamed R, Turbide C, Buret AG, Heitman SJ. Infection control in ERCP using a duodenoscope with a disposable cap (ICECAP): rationale for and design of a randomized controlled trial. BMC Gastroenterol. 2020 Mar 12;20(1):64. doi: 10.1186/s12876-020-01200-7. PMID 32164535